CLINICAL TRIAL: NCT03110705
Title: Recreational Diving Practice for Stress Management: an Exploratory Controlled Trial
Brief Title: Recreational Diving Practice for Stress Management
Acronym: DIVSTRESS
Status: Completed | Type: Observational
Sponsor: Institut de Recherche Biomedicale des Armees (Other Government)
Responsible Party: Principal Investigator, Marion Trousselard, senior research, Institut de Recherche Biomedicale des Armees
Other Study IDs: 2015-A00133-46
Record Dates: First submitted 2017-03-18; First posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Psychological Stresses
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- recreational diving group: middle-class populations registered at a leisure sports club
  Interventions: Behavioral: sport
- recrational multisport course: middle-class populations registered at a leisure sports club
  Interventions: Behavioral: sport

INTERVENTIONS:
Behavioral: sport — recreaational sport : diving or multisport

SUMMARY:
Within the components of Scuba diving there are similarities with meditation and mindfulness techniques. Perceived stress is known to be diminished during meditation practice. This study evaluates the benefits of scuba diving on perceived stress and mindful functioning.

DETAILED DESCRIPTION:
Background: within the components of Scuba diving there are similarities with meditation and mindfulness techniques. Perceived stress is known to be diminished during meditation practice. This study evaluates the benefits of scuba diving on perceived stress and mindful functioning.

Method: A recreational diving group, composed of 37 subjects, was compared with a multisport control group, composed of 30 subjetcs, on perceived stress, mood, well-being and mindfulness by answering auto-questionnaires before and after a one-week long course. For the diving group, stability of the effects was evaluated one month later using similar auto-questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* More than 18
* registered at a leisure sports club

Exclusion Criteria:

* they were undergoing medical treatment for psychological issues at the time of the study
* they had taken part in a stress management program prior to recruitment for the current study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: middle-class populations registered at a leisure sports club were included: one population sample registered for a one-week recreational scuba diving course (37 subjects, diving group) and one population sample registered for a one-week multisport course (30 subjects, control group).
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2015-03-12 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2016-11-17 (Actual)

PRIMARY OUTCOMES:
perceived stress | change from baseline after one week sport (e.g. baseline and one week)
  questionnaire

SECONDARY OUTCOMES:
mindfulness | change from baseline after after one week sport (e.g. baseline and one week)
  questionnaire

IPD SHARING:
Plan to Share IPD: No